CLINICAL TRIAL: NCT01300754
Title: Phase 2 Study of Dextrose Injection for Sport-Limiting Osgood Schlatter Disease in Adolescents.
Brief Title: Effectiveness of Dextrose Injection for Osgood-Schlatter Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad Nacional de Rosario (Other)
Responsible Party: Gastón Andrés Topol, M.D., Hospital Provincial de Rosario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNRosario
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-01

CONDITIONS: Osgood-Schlatter Disease
Keywords: Osgood-Schlatter; Tendinosis; Apophysitis; Enthesopathy; Dextrose.
MeSH Terms: conditions — Osteochondrosis; Tendinopathy; Enthesopathy | interventions — Glucose; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dextrose (Active Comparator)
  Interventions: Procedure: Dextrose Injection
- Lidocaine (Active Comparator)
  Interventions: Procedure: Lidocaine Injection
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Procedure: Dextrose Injection — 12.5 Dextrose in 1% Lidocaine injected monthly for 3 months with a 27 gauge needle on painful areas of the tibial tuberosity, under the patellar tendon.
  Arms: Dextrose
Procedure: Lidocaine Injection — 1% Lidocaine injected monthly for 3 months with a 27 gauge needle on painful areas of the tibial tuberosity, under the patellar tendon.
  Arms: Lidocaine
Other: Usual Care — Therapist supervised exercises that are standard of care for Osgood-Schatter Disease as well as relative rest and gradual resumption of pain-limited sport.
  Arms: Usual Care

SUMMARY:
Objective: To examine the potential of dextrose injection versus lidocaine injection versus supervised usual care to change pain/function/activity levels in adolescent athletes with Osgood-Schlatter Disease (OSD).

DETAILED DESCRIPTION:
Patients and methods: Girls ages 9-15 years old and boys ages 10-17 years old will be assigned to either therapist-supervised usual care, or to double-blind injection of 1% lidocaine solution with or without 12.5% dextrose. Injections will be administered monthly for three months. All subjects will then be offered dextrose injections monthly as needed. Change in the Nirschl Pain Phase Scale (NPPS) will serve as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Age:9-15 year old girls and 10-17 year old boys
* Pain Location: Anterior knee.
* Sport Type: Jumping or kicking sport.
* Team Member with Coach: Member of and organized team with a coach.
* Imitation of exact pain and precise location to the tibial tuberosity with a single leg squat.
* At least 2 months of formal and gently progressive hamstring stretching, quads strengthening, and gradual sports reintroduction.
* Pain with sport at least 3 months.

Exclusion Criteria:

* Patellofemoral crepitus
* Patellar origin tenderness

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaston A Topol, Dr., Principal Investigator — Hospital Provincial de Rosario
Locations (1):
- Hospital Provincial de Rosario, Rosario, Santa Fe Province, Argentina

REFERENCES:
- [Derived] Topol GA, Podesta LA, Reeves KD, Raya MF, Fullerton BD, Yeh HW. Hyperosmolar dextrose injection for recalcitrant Osgood-Schlatter disease. Pediatrics. 2011 Nov;128(5):e1121-8. doi: 10.1542/peds.2010-1931. Epub 2011 Oct 3. PMID 21969284